CLINICAL TRIAL: NCT05611801
Title: AN OPEN-LABEL STUDY IN PEDIATRIC (<18 YEARS OF AGE), SEVERE HEMOPHILIA A PARTICIPANTS (COAGULATION FACTOR ACTIVITY <1%) WITH OR WITHOUT INHIBITORS OR MODERATELY SEVERE TO SEVERE HEMOPHILIA B PARTICIPANTS (COAGULATION FACTOR ACTIVITY =2%) WITH OR WITHOUT INHIBITORS COMPARING 12 MONTHS OF HISTORICAL STANDARD TREATMENT TO MARSTACIMAB PROPHYLAXIS
Brief Title: A Clinical Trial of Study Medicine (Marstacimab) in Pediatric Patients With Hemophilia A or Hemophilia B
Acronym: BASIS KIDS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7841008; ANTI-TFPI PEDIATRIC STUDY (Other: Alias Study Number); 2022-500495-65-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-10-27; First posted 2022-11-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Factor VIII Inhibitor; Factor IX Inhibitor; PF-06741086; Marstacimab; Anti-TFPI; Factor VIII; Factor IX; Inhibitors; Anti-Tissue Factor Pathway Inhibitor (TFPI); Subcutaneous (sc); Prophylaxis; On-Demand; BASIS KIDS; Inhibitor; SC; Subcutaneous; Injection; On demand; aTFPI; Severe hemophilia; Severe bleeding; Hemophilia
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Hemorrhage | interventions — marstacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- marstacimab (PF-06741086) (Experimental): Weekly subcutaneous injections.
  Interventions: Drug: marstacimab

INTERVENTIONS:
Drug: marstacimab — marstacimab
  Other Names: PF-06741086

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called marstacimab) for the potential treatment of hemophilia in pediatric patients.

This study will enroll pediatric participants from ages 1 to 17 years in a sequential manner. The study will open enrollment to adolescent participants aged 12 to 17 years first. Then children aged 6 to 11 years will be permitted to enroll. Lastly, children aged 1 to 5 years will be permitted to enroll.

This study will enroll participants who:

* have severe Hemophilia A or moderately severe to severe Hemophilia B (with or without inhibitors)
* have accurate historical records documenting all factor VIII, factor IX, or bypass agent infusions and hemophilia bleed events for at least 1 year prior to entering the study
* if a non-inhibitor patient, must be on a stable routine prophylaxis regimen with factor VIII or factor IX replacement products for at least 12 months prior to study entry
* if an inhibitor patient, must be on an on-demand bypass treatment regimen during the 12 months prior to study entry

All participants in this study will receive marstacimab to use prophylactically. Marstacimab will be given once a week as a subcutaneous (under the skin) shot. The first dose of marstacimab will be given at the study site by the study site staff. During the 12-month treatment period, weekly doses of marstacimab can be given at home, or if preferred, the doses may be given by the study site staff.

To help us determine if the study medicine is safe and effective, we will compare participant experiences when they are taking the study medicine to a historical period when they were not. Researchers want to see if the study medicine works to prevent the bleeding episodes commonly experienced by patients with Hemophilia.

Participants will be in this study for about 14 months (approximately 1 month in a Screening period, 12 months receiving treatment, and 1 month in a follow-up period) during which they will visit the study site at least 10 times. If preferred, and if local regulations allow it, 2 of the study visits can be completed at the participant's home instead of at the study site. There will also be 6 scheduled telephone calls approximately every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Male participants of appropriate age and required minimum weight
* Participants aged 12 to 17 years must be at least 25 kgs at time of consent.
* Participants aged 6 to 11 years must be at least 19 kgs at time of consent.
* Minimum weight requirement for participants aged 1 to 5 years is to be determined.
* Participants with a diagnosis of severe hemophilia A or moderately severe to severe hemophilia B
* Participants must have at least 1 year of diary and/or medical records available in which exogenous FVIII or FIX replacement or bypass agent infusions and hemophilic bleeding episodes were consistently documented over the 12 months prior to the time of consent.

Participants who are enrolled into the Non-Inhibitor Cohort must also meet the following criteria:

* No current detectable inhibitor and no documented history of inhibitors in the 5 years prior to consent
* Must have at least 50 exposure days to FVIII/FIX replacement products
* Must be at least 80% compliant with a stable and effective routine prophylaxis regimen with FVIII/FIX replacement products, for at least 12 months prior to consent

Participants who are enrolled into the Inhibitor Cohort must also meet the following criteria:

* Documentation of current high titer inhibitor (≥5 BU/mL); or current low titer inhibitor (<5 BU/mL) refractory to FVIII or FIX replacement and with FVIII or FIX recovery <60% of expected within previous 12 months prior to the time of consent
* Participants who have documented inhibitors while on factor-replacement therapy but who do not meet the high quantitative inhibitor criteria described in the prior bullet at the time of screening (eg, participant with a previously documented high-titer inhibitor ≥5 BU/mL) and whose condition precludes re-challenge with FVIII or FIX replacement may be considered for eligibility on a case-by-case basis with discussion and agreement from the Pfizer medical monitor.
* Hemophilia A participants with on-demand treatment regimen with ≥12 bleeding episodes or hemophilia B participants with on-demand treatment regimen with ≥8 bleeding episodes (spontaneous or traumatic) necessitating treatment with bypass factor in the 12 months prior to informed consent
* Participants must be on an on-demand bypass treatment regimen during the 12 months prior to informed consent

Exclusion Criteria:

* Known coronary artery, thrombotic, or ischemic disease, or current evidence of congenital or acquired thrombophilic disease such as Anti-thrombin III deficiency, Factor V Leiden mutation, prothrombin 20210 mutation, protein C deficiency, protein S deficiency and antiphospholipid syndrome.
* Known planned surgical procedure during the planned study period
* Known hemostatic defect other than hemophilia A or B
* Abnormal hematology, renal or hepatic function laboratory results at screening
* Other acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator
* Individuals with known allergic reaction or hypersensitivity to hamster protein or other components of the study intervention
* Current routine prophylaxis with bypassing agent, non-coagulation non-factor replacement therapy (eg, emicizumab), or any previous treatment with a gene therapy product for treatment of hemophilia
* Participants with inhibitors who are being treated using a prophylaxis treatment regimen with a bypass agent, and, participants who have previously received non-factor-based hemophilia therapy (eg, fitusiran, concizumab, emicizumab) will be considered on a case-by-case basis, only after discussion and agreement between the investigator and the Pfizer medical monitor
* Regular use of immunomodulatory medications (eg, IVIG, routine systemic corticosteroids, rituximab)
* Use of systemic antifibrinolytics, medications that may increase the risk of bleeding, and certain non-steroidal anti-inflammatory drugs within 120 hours of first dose of study intervention and while on study
* Ongoing or planned use of ITI, or prophylaxis with FVIII or FIX replacement at any time after initiation of treatment with study intervention
* Participation in other studies involving investigational drug(s) or investigational vaccine(s) within 30 days (or as determined by local requirements) or 5 half-lives prior to study entry or during study participation
* Previous exposure to marstacimab during participation in other marstacimab clinical studies
* CD4 cell count ≤200/uL if HIV-positive
* Abnormal ECG of clinical relevance that may affect participant safety or interpretation of study results
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members

Ages: 1 Year to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2028-09-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Annualized bleeding rate (ABR) of treated bleeding events | Baseline to end of 12-month treatment period
  Derived for each subject for each period (historical and study treatment) by using the following formula: ABR = number of bleeds requiring treatments/ (days on treatment period / 365.25)
Incidence of adverse events and serious adverse events | Screening through end of follow-up period (approximately 14 months)
Incidence and severity of thrombotic events | Baseline to end of 12-month treatment period
Incidence and severity of thrombotic microangiopathy | Baseline to end of 12-month treatment period
Incidence and severity of disseminated intravascular coagulation/consumption coagulopathy events | Baseline to end of 12-month treatment period
Immunogenicity (incidence of ADA and clinically significant persistent NAb against marstacimab) | Baseline to end of 12-month treatment period
Incidence and severity of injection site reaction | Baseline to end of 12-month treatment period
Incidence of severe hypersensitivity and anaphylactic reactions | Baseline to end of 12-month treatment period

SECONDARY OUTCOMES:
Incidence of joint bleeds (treated) | Baseline to end of 12-month treatment period
Incidence of spontaneous bleeds (treated) | Baseline to end of 12-month treatment period
Incidence of target joint bleeds (treated) | Baseline to end of 12-month treatment period
Incidence of total bleeds (treated and untreated) | Baseline to end of 12-month treatment period
Number of target joints | Baseline to end of 12-month treatment period
Change from baseline in joint health as measured by the HJHS for participants ≥4 years of age | Baseline to end of 12-month treatment period
Changes in quality of life measured by Haem-A-QoL/Haemo-QoL (using age-dependent versions for participants ≥8 years of age) | Baseline to end of 12-month treatment period
Changes in quality of life measured by pedHAL (using age-dependent versions for participants ≥4 years of age) | Baseline to end of 12-month treatment period
Changes in quality of life measured by Patient Global Impression of Change - Hemophilia for participants ≥4 years of age | Baseline to end of 12-month treatment period
Changes in quality of life measured by Health Utilities Measure (EQ-5D-Y) for participants ≥4 years of age | Baseline to end of 12-month treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- Intermountain - Primary Children's Hospital, Salt Lake City, Utah, United States
- Arbesu Hematología, Mendoza, Argentina
- Australia (2):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal Children's Hospital, Melbourne, Victoria
- Medizinische Universität Wien, Vienna, Vienna, Austria
- HEMOES, Vitória, Espírito Santo, Brazil
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Hamilton Health Sciences - McMaster University Medical Centre, Hamilton, Ontario/canada
- China (7):
  - Beijing Children's hospital, Capital Medical University, Beijing, Beijing Municipality
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College of HUST/Pediatric Hematology Department Pharmacy, Wuhan, Hubei
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Institute of hematology&blood disease hospital, Tianjin, Tianjin Municipality
- Detska nemocnice FN Brno, Brno, Brno-město, Czechia
- Denmark (2):
  - Rigshospitalet, Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland
- Hôpital Universitaire Necker Enfants Malades, Paris, France
- Charité Campus Virchow-Klinikum, Berlin, Germany
- India (3):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - K.J. Somaiya Hospital, Mumbai, Maharashtra
  - Nil Ratan Sircar Medical College and Hospital, Kolkata, West Bengal
- Sheba Medical Center, Ramat Gan, Central District, Israel
- Italy (5):
  - IRCCS Istituto Giannina Gaslini, Genoa, Liguria
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Ospedale Pediatrico Bambino Gesù IRCCS, Rome, ROMA
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
- Japan (5):
  - Hyogo prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - Nagano Children's Hospital, Azumino, Nagano
  - Nara Medical University Hospital, Kashihara, Nara
  - Saitama Prefectural Children's Medical Center, Saitama-shi, Saitama
  - Saga University Hospital, Saga
- Arké SMO S.A de C.V, Veracruz, Mexico
- Saudi Arabia (2):
  - King Fahad Specialist Hospital - Dammam, Dammam, Eastern Province
  - King Faisal Specialist Hospital & Research Center, An Narjis
- Slovakia (2):
  - Detska fakultna nemocnica Kosice, Košice
  - Univerzitna nemocnica Martin, Martin
- South Africa (2):
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
- South Korea (3):
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyung Hee University Hospital at Gangdong, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Hospital, Daegu, Taegu-kwangyǒkshi
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (3):
  - Changhua Christian Hospital, Changhua County, Changhua
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (7):
  - Istanbul Universitesi Istanbul Tıp Fakultesi Hastanesi, Istanbul, İ̇stanbul
  - Ege Universitesi Hastanesi, Izmir, İ̇zmir
  - Erciyes University, Talas, Kayseri
  - Acibadem Adana Hospital, Adana
  - Gazi University Health Research and Application Center Gazi Hospital, Ankara
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri, Kayseri
  - Ondokuz Mayıs Universitesi, Samsun
- United Kingdom (4):
  - Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Birmingham Children's Hospital, Birmingham
  - Evelina London Children's Hospital, London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7841008